CLINICAL TRIAL: NCT00981890
Title: A Phase I Study of Stereotactic Radiosurgery Concurrent With Sunitinib in Patients With Brain Metastases
Brief Title: Stereotactic Radiosurgery With Sunitinib for Brain Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 09-0115-C
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Brain Metastases
Keywords: Brain Metastases; Stereotactic radiosurgery; Sunitinib; Patients with Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib is a tablet that is taken by mouth every day. Patients will be treated with Sunitinib alone for 7 days. On the seventh day of taking the drug they will be given SRS. Sunitinib will continue for seven days per week after SRS, and depending on how far along the study is when patients join, they may continue taking the drug for up to 13 weeks after SRS.

SUMMARY:
The purpose of this study is to determine the maximum dose of sunitinib that can be tolerated when treatment is combined with radiotherapy. Patients who decide to take part in the study will start taking sunitinib alone for 7 days. On the seventh day of taking sunitinib, patients will be given stereotactic radiosurgery (SRS).

The dose of radiation that patients will receive when they are given SRS is a standard dose used to help shrink brain metastases. The dose of radiation and the way it is delivered is not experimental.

Patients will then continue to take sunitinib seven days per week after SRS, and depending on how far along the study is when they join, they may continue taking the drug for up to 13 weeks after SRS. Patients will undergo weekly assessment during study treatment.

DETAILED DESCRIPTION:
Brain metastases occur in 20% to 40% of all patients with cancer, with an incidence 10 times higher than that of primary malignant brain tumours. The reported median survival of patients with brain metastases is only 1-2 months with corticosteroids and 5-7 months with whole brain radiotherapy (WBRT). But with improvements in neuroimaging, brain metastases are being diagnosed more frequently and with a lower burden of disease, such that approximately 50-60% of patients have 1 to 4 brain metastases at diagnosis. In these patients, stereotactic radiosurgery (SRS), a single high dose of radiation delivered with high precision to the target lesion, is being used increasingly as an alternative to surgical resection or as an adjunct to WBRT. The addition of SRS to WBRT has provided improvements in local control and functional autonomy for patients with oligometastatic brain disease, supporting the hypothesis that SRS increases efficacy against tumours resistant to the significantly lower doses used in WBRT.

SRS can accomplish destruction of a defined intracranial target through precise targeting of a high dose of radiation with a sharp dose fall off at the target boundaries and minimal damage to surrounding tissue. Brain metastases are well suited for SRS as they are often small, radiographically well-circumscribed, pseudo-spherical tumors that are non-infiltrative, and they are often located at the gray-white junction, where toxicity to critical structures is minimal. SRS toxicity is low (<5%).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven malignancy (original biopsy is adequate as long as the brain imaging is consistent with brain metastases).
* Patients age 18 years of age or older, as the effects of Sunitinib at the recommended therapeutic dose are unknown in children.
* A contrast-enhanced MRI demonstrating the presence of 1-3 brain metastases performed within four weeks prior to registration.
* The dominant contrast-enhancing intraparenchymal brain metastases must be well-circumscribed and must have a maximal diameter of ≤ 4.0 cm in any direction on the enhanced scan. If multiple lesions are present and one lesion is at the maximum diameter, the other(s) must not exceed 3.0cm in maximum diameter.
* Life expectancy > 3 months
* RPA Class 1 and RPA Class 2 patients with stable primary disease
* No systemic anti-cancer therapy within 30 days of starting or completing study treatment
* Patients must have normal organ and marrow function as defined in the protocol.
* Effects of Sunitinib on the developing human fetus at the recommended therapeutic dose are unknown. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with leptomeningeal metastases documented by MRI or CSF evaluation
* Evidence of intratumoural or peritumoural hemorrhage deemed significant by the treating physician
* Patients with metastases within 5 mm of the optic chiasm or optic nerve
* Patients with metastases in the brainstem (midbrain, pons, or medulla).
* < 4 weeks since any major surgery. (Previous brain surgery, including craniotomy for tumour resection [except cerebral metastases] or biopsy is permissible.)
* Prior resection of cerebral metastasis
* Previous cranial radiation. Patients may have had radiation therapy to other anatomical sites, but must have recovered from acute toxic effects prior to registration. At least 2 weeks must have elapsed since last dose of radiation before registration.
* Treatment with a non-approved or investigational drug concurrently or within 30 days before Day 0 of study treatment or within 30 days after the last day of study treatment.
* Treatment with sunitinib or other inhibitors of the VEGF signalling axis within 30 days before Day ) of study treatment or within 30 days after last day of study treatment.
* Bleeding disorders.
* Thrombolytic therapy within 4 weeks
* Concurrent use of anticoagulant or antiplatelet drugs
* Concurrent use of enzyme-inducing anti-epileptic drugs
* Patients with any condition that impairs their ability to swallow Sunitinib (e.g. gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with poorly controlled hypertension (systolic blood pressure of 150 mmHg or higher, or diastolic blood pressure of 100 mmHg or higher) are ineligible
* New York Heart Association (NYHA) Class III or IV disease
* NYHA class II disease controlled with treatment and monitoring allowed
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Sunitinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Pregnant women. These patients are excluded because there is an unknown but potential risk for adverse events in the fetus. Because there is also an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Sunitinib. Breastfeeding should be discontinued if the mother is treated with Sunitinib.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Sunitinib.
* Individuals with MRI non-compatible metal in the body, or unable to undergo MRI procedures.
* Allergy to gadolinium
* Allergy to Iodine Contrast Agent
* Glomerular Filtration Rate of less than 30ml.min/1.73m2 as measured by creatinine clearance through the Cockcroft-Gault formula [(140-age) X Mass in kg / 72 X plasma creatinine (mg/dl)]
* Primary germ cell tumor, small cell carcinoma, or lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Determine the safety and maximum tolerated dose of Sunitinib when combined concurrently with SRS in patients with 1-3 brain metastases | 2 years

SECONDARY OUTCOMES:
Assess: late toxicities/Tx effect on cognitive function/potential prognostic factors/time to Intracranial Local & Distant Progression/brain Progression-free Survival/alterations in tumour perfusion parameters & effects in normal brain tissue | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Chung, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada